CLINICAL TRIAL: NCT03304899
Title: Early Fibrinogen Concentrate in Isolated Traumatic Brain Injury and the Effect on Post Bleeding & Complications
Brief Title: Fibrinogen Concentrate in Isolated Traumatic Brain Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leila Dehghani (Other)
Responsible Party: Sponsor-Investigator, Leila Dehghani, Early fibrinogen concentrate in severe isolated traumatic brain injury and the effect on post bleeding and complications., Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Isfahan University
Record Dates: First submitted 2017-09-09; First posted 2017-10-09 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Traumatic Brain Injury; Hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case group (Experimental): Severe isolated Traumatic Brain injury patients with serum fibrinogen level under 200 mg/dl that receive Fibrinogen concentrate after common emergency resuscitation. Instruction:
  1. Airway control & breathing.
  2. Circulation (Serum therapy, Epinephrine,Packed cell, FFP and ...).
  3. Fibrinogen Concentrate(IV injection): Each vial contains 1gr fibrinogen concentrate. Fibrinogen concentrate will be given until serum fibrinogen level riches to 200 mg/dl.
  Dose (mg/kg body weight) = ([Target level (mg/dL) - measured level (mg/dL)])/(1.7 (mg/dL per mg/kg body weight))
  Interventions: Drug: RiaSTAP Injectable Product
- Control group (Active Comparator): Severe isolated Traumatic Brain injury patients with serum fibrinogen level under 200 mg/dl that receive common emergency resuscitation. Instruction:
  1. Airway control & breathing.
  2. Circulation (Serum therapy, Epinephrine,Packed cell, FFP and ...).
  Interventions: Drug: RiaSTAP Injectable Product

INTERVENTIONS:
Drug: RiaSTAP Injectable Product — RiaSTAP, Fibrinogen Concentrate (Human) is a human blood coagulation factor indicated for the treatment of acute bleeding episodes.
  Dose (mg/kg body weight) =
  ([Target level (mg/dL) - measured level (mg/dL)])/(1.7 (mg/dL per mg/kg body weight))

SUMMARY:
Fibrinogen is a unique precursor of fibrin and cannot be compensated for by other coagulation factors. If plasma fibrinogen concentrations are insufficient, hemostatic clots cannot be formed with the appropriate firmness. In severe traumatic brain injury(TBI) patients, plasma fibrinogen concentrations decrease earlier and more frequently than other coagulation factors,predicting massive bleeding and death.

The purpose of this study is to try early injection of fibrinogen concentrate in severe isolated traumatic brain injury and investigation the effect of it on post bleeding and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe isolated traumatic brain injury.

Exclusion Criteria:

* Severe abdomen or extremities trauma.
* Severe bleeding from abdomen or extremities.
* Congenital coagulopathy (Hemophilia, protein S and C deficiency, Factor 5 Leiden deficiency and ...).
* Warfarin, Heparin, Enoxaparin, Dabigatran and other anticoagulation drugs consumption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-12-21 (Estimated); Study Completion 2020-01-21 (Estimated)

PRIMARY OUTCOMES:
Mortality rate. | Until 90 days after admission.
  Mortality rate after injection of fibrinogen concentrate.
Average of serum fibrinogen level. | Immediately after admission.
  Average of serum fibrinogen level in iTBI patient.
The effect of early fibrinogen on post trauma bleeding (Intracranial hemorrhage). | 2, 6, 24, 72 hours and 30 , 90 days after admission.
  The need to packed cell, FFP, Platelete.

SECONDARY OUTCOMES:
The complications that related to fibrinogen concentrate. | until 90 days after admission.
  like DVT, PTE, MI.by measurement of serum D-dimer for DVT and PTE and serum Troponin C for MI.

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan university of medical science., Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided